CLINICAL TRIAL: NCT06412770
Title: Director, World Health Organization (WHO)
Brief Title: Effect of Tai Chi on Symptoms in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, qinxiu zhang, professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: chengduTCM20240314
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Dialysis; Complications; Chinese Medicine; Quality of Life
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi intervention group (Experimental): Tai Chi intervention group
  Interventions: Behavioral: Tai chi
- Tai Chi Imagery Intervention Group (Placebo Comparator): Tai Chi Imagery Intervention Group
  Interventions: Behavioral: Tai Chi imagery
- Control group (Other): no intervention
  Interventions: Other: no-intervention

INTERVENTIONS:
Behavioral: Tai chi — Participants will be asked to do Tai Chi for 30 minutes three times a week
  Arms: Tai Chi intervention group
Behavioral: Tai Chi imagery — Participants will be asked to do Tai Chi imagery for 30 minutes three times a week
  Arms: Tai Chi Imagery Intervention Group
Other: no-intervention — The comparison group will be given usual care
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn about the effect of Tai Chi on symptoms in hemodialysis patients.The main question[s] it aims to answer are: the effect of Tai Chi on symptoms or the quality of life in hemodialysis patients .Participants will be divided into three groups, one group will be asked to do Tai Chi for 30 minutes three times a week, and the other group will be asked to do Tai Chi imagery for 30 minutes three times a week. The comparison group will be given usual care. Researchers will compare the efficacy of symptoms and quality of life in dialysis patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18;
* Dialysis age≥ 3 months;
* Survival≥ 12 months;
* The patient has the ability to move independently, can learn independently, and has no reading and comprehension disabilities;
* Informed consent

Exclusion Criteria:

* Inability to move autonomously;
* Have a mental disorder;
* Other serious complications occur

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of life quality after treatment | Assessment was performed at 4, 8, and 12 weeks after treatment
  The effects of tai Chi on symptoms (fatigue, pain, depression, sleep) of hemodialysis patients were assessed by scale